CLINICAL TRIAL: NCT02887534
Title: A Randomized, Double-blind, Active and Placebo-controlled, Study of SPARC1401 in Subjects With Moderate to Severe Acute Low Back Pain
Brief Title: Evaluation of Efficacy and Safety of SPARC1401 in Acute Low Back Pain
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharma Advanced Research Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CLR_14_01
Record Dates: First submitted 2016-07-20; First posted 2016-09-02 (Estimated); Last update posted 2019-05-03 (Actual); Status verified 2019-05

CONDITIONS: Acute Muscle Pain
MeSH Terms: interventions — tizanidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm 1 (Experimental): three times medication; SPARC1401-low dose
  Interventions: Drug: SPARC1401-low dose; Drug: Placebo1401
- Arm 2 (Experimental): three times medication; SPARC1401-mid dose
  Interventions: Drug: SPARC1401-mid dose; Drug: Placebo1401
- Arm 3 (Experimental): three times medication; SPARC1401-high dose
  Interventions: Drug: SPARC1401-high dose; Drug: Placebo1401
- Active comparator (Active Comparator): Reference1401; To be administered 3 times a day
  Interventions: Drug: Reference1401 (Tizanidine)
- Arm 5 (Placebo Comparator): Placebo1401 - 3 three times a day
  Interventions: Drug: Placebo1401

INTERVENTIONS:
Drug: SPARC1401-low dose — SPARC1401- low dose
  Other Names: Test 1
  Arms: Arm 1
Drug: SPARC1401-mid dose — SPARC1401- mid dose
  Other Names: Test 2
  Arms: Arm 2
Drug: SPARC1401-high dose — SPARC1401-high dose
  Other Names: Test 3
  Arms: Arm 3
Drug: Reference1401 (Tizanidine) — Reference1401 (Tizanidine) three times a day
  Other Names: Reference1401
  Arms: Active comparator
Drug: Placebo1401 — Placebo
  Other Names: Placebo intervention
  Arms: Arm 1; Arm 2; Arm 3; Arm 5

SUMMARY:
A phase 2 randomized clinical trial to evaluate efficacy and safety of SPARC1401 at three dose levels in patients with acute low back pain

ELIGIBILITY:
Inclusion Criteria:

* Gives informed and written consent and is able to comply with all study assessments scheduled in the protocol
* Males or females aged 18 to 80 years (inclusive).
* Female subjects should be surgically sterile (bilateral tubal ligation at least 6 months prior to randomization, bilateral oophorectomy or hysterectomy performed) or if they are of child-bearing potential, should be willing to practice an acceptable method of birth control from screening to completion of study.
* Subjects will be considered eligible for this trial based on medical evaluation, electrocardiogram and laboratory values at screening, and laboratory values outside normal range considered of no clinical significance by the investigator

Exclusion Criteria:

* History or presence of clinically significant or uncontrolled cardiovascular, respiratory, neurological, psychiatric, hepatic, renal, gastrointestinal, hematological, or sleep disorder
* History or clinical signs or symptoms suggestive of stenosing peptic ulcer, pyloroduodenal obstruction, or inflammatory bowel disease
* History of diagnosis of cancer within 5 years prior to screening
* History of narrow-angle glaucoma, symptomatic prostatic hypertrophy, or bladder-neck obstruction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-11 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Rating for medication helpfulness on five point scale: 0 - poor, 1 - fair, 2 - good, 3 - very good, 4 - excellent | Day 4

SECONDARY OUTCOMES:
Rating for medication helpfulness on five point scale: 0 - poor, 1 - fair, 2 - good, 3 - very, 4 - excellent | Day 8

IPD SHARING:
Plan to Share IPD: No